CLINICAL TRIAL: NCT04128774
Title: The Function and Composition of B Cells in Participants With Glioblastoma Treated With and Without Dexamethasone
Brief Title: Function and Composition of Regulatory B Cells in Participants With Glioblastoma
Acronym: GBMdexaB
Status: Terminated | Type: Observational
Why Stopped: To few participants
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Mathilde Kouwenhoven, Neurologist, Amsterdam UMC, location VUmc
Other Study IDs: 2019.554; CCA2018-5-50 (Other Grant/Funding Number: Cancer Center Amsterdam Research Foundation); NL71359.029.19 (Registry Identifier: Nederlands Trial Register)
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma, Adult
Keywords: Glioma; Glioblastoma; Adult; Dexamethasone; B cells; Regulatory B cells
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GBM-dexa: Participants with clinical diagnosis of GBM, that require dexamethasone due to neurological deficits. Dose is based on the clinical judgement of the treating physician but should be given at least two weeks. Dexamethasone is given once a day.
  Interventions: Drug: Dexamethasone
- GBM-control: Participants with clinical diagnosis of GBM not requiring dexamethasone treatment.

INTERVENTIONS:
Drug: Dexamethasone — The case group receives dexamethasone based on the clinical indication.
  Other Names: Dexamethasone indicated based on the clinical indication.
  Groups: GBM-dexa

SUMMARY:
Rationale: This project elaborates on a novel finding of the investigators that has not yet been reported in literature, namely the presence of elevated levels of atypical B cells in participants with glioblastoma. ln the period 2015 2018 the investigators analysed the blood immune subset composition of a cohort of 180 participants undergoing neurosurgery. The most relevant finding was the presence of an abnormally elevated level of B cells in the blood of the great majority of participants with glioblastoma. These B cells may be involved in the immunosuppression associated with glioblastoma that makes this tumor refractory to immunotherapy. Multiple regression analysis indicated that the increase in the frequency of atypical B cells in participants' peripheral blood was related with the administration of dexamethasone prior to surgery. However, this study design did not allow the investigators to address the causality of the relationship between dexamethasone and atypic B cell dysregulation. Alternative treatments to dexamethasone exist.

Objective: To investigate the effect of dexamethasone in the dysregulation of atypic B cells in participants with glioblastoma.

Study design: Observational case control pilot study with 20 participants (10 per group).

Study population: Newly diagnosed participants with glioblastoma. Intervention (if applicable): Observational study. Main study parameters/endpoints: Changes in the immune subset composition and functionality in the peripheral blood of participants with glioblastoma upon administration of dexamethasone for neurological signs of peritumoral edema (oral dexamethasone).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The investigators will collect blood (28 ml) during the first visit and again (28 ml) at the time of surgery (2 weeks ± 3 days). There will not be additional site visits, physical examinations or any other tests, questionnaires. Blood collection is only a minor discomfort and it does not represent any additional risk.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis Glioblastoma Patients are 18 years or older at first diagnosis

Exclusion Criteria:

No indication for surgery to confirm radiological diagnosis Not able or willing to give informed consent Allergy or intolerance to dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis Gliobastoma
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Frequency of regulatory B cells in blood of participant with Glioblastoma | Two weeks
  ldentify if dexamethasone treatment alters the frequency and functionality of atypic B cells (CD25+CD95Fas+-B cells) in blood in GBM.

SECONDARY OUTCOMES:
Changes in frequency of regulatory B cells after treatment of participants with Glioblastoma with dexamethasone | Two weeks
  Changes in the frequency and functionality of regulatory B cells in blood after two weeks of treatment with dexamethasone.
Changes in frequency of regulatory B cells in participants with Glioblastoma | Two weeks
  Changes in the frequency and functionality of regulatory B cells in blood in patients not treated with dexamethasone.

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde CM Kouwenhoven, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam Medical Universities, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data will be stored in coded form in a Castor database. At this moment data will not be available to other researchers.

REFERENCES:
- [Background] Dusoswa SA, Verhoeff J, Garcia-Vallejo JJ. OMIP-054: Broad Immune Phenotyping of Innate and Adaptive Leukocytes in the Brain, Spleen, and Bone Marrow of an Orthotopic Murine Glioblastoma Model by Mass Cytometry. Cytometry A. 2019 Apr;95(4):422-426. doi: 10.1002/cyto.a.23725. Epub 2019 Jan 31. PMID 30701669